CLINICAL TRIAL: NCT03773731
Title: Impact of High Intensity Interval Training vs. Continuous Aerobic Training on Platelet Insulin Resistance, Platelet Function and Hepatic Steatosis in Patients With Prediabetes
Brief Title: High Intensity Interval Training in Prediabetes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical University of Vienna (Other)
Collaborators: University of Vienna, Institute for Sport Science (Unknown); Sanatorium Hera Vienna (Unknown)
Responsible Party: Principal Investigator, Stefan Heber, Dr.med.univ. Dr.rer.nat., Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: Exercise_platelet_insulin
Record Dates: First submitted 2018-12-10; First posted 2018-12-12 (Actual); Last update posted 2019-01-09 (Actual); Status verified 2019-01

CONDITIONS: Prediabetic State
MeSH Terms: conditions — Prediabetic State | interventions — High-Intensity Interval Training

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High intensity interval training (Experimental): 3x/week the following 45 min training protocol on bicycle ergometer for 12 weeks:
  * 5 minutes warm-up phase with a power output of 40% of the maximal power output achieved in an incremental exercise test
  * 30 minutes: intensive cycling bouts of 60s interspersed with 60s of recovery intervals. Power output will be 90% (week 1-6) or 95% (week 7-12) of the maximal power output of the exercise test during the intensive cycling bouts. During recovery intervals, subjects will pedal with a power output of 30% (week 1-6) or 35% (week 7-12) of the maximal power output of the exercise test.
  * 10 minutes with 30% of maximal power output.
  Interventions: Behavioral: High intensity interval training (HIIT)
- Moderate intensity continuous training (Active Comparator): 3x/week the following 45 min training protocol on bicycle ergometer for 12 weeks:
  * 5 minutes warm-up phase with a power output of 40% of the maximal power output achieved in an incremental exercise test
  * 30 minutes: Continuous training with 60% (week 1-6) or 65% (week 7-12) of maximal power output
  * 10 minutes with 30% of maximal power output.
  Interventions: Behavioral: Moderate intensity continuous training (MICT)

INTERVENTIONS:
Behavioral: High intensity interval training (HIIT) — Exercise training on bicycle ergometer with high intensity bouts of 1 min interspersed by low intensity recovery intervals
  Arms: High intensity interval training
Behavioral: Moderate intensity continuous training (MICT) — Exercise training on bicycle ergometer with moderate intensity (60 - 65 % of individual maximal power output)
  Arms: Moderate intensity continuous training

SUMMARY:
This trial investigates if high intensity interval training is more effective than moderate intensity continuous training in suppressing platelet reactivity and hepatic fat content in prediabetic individuals.

DETAILED DESCRIPTION:
Background:

The prevalence of type 2 diabetes mellitus (T2DM) is rising dramatically. T2DM represents a major cause for cardiovascular disease -related mortality and morbidity and increasingly burdens healthcare systems. While the fundamental pathomechanism of T2DM is insulin resistance of muscle and adipose tissue, recent studies demonstrate that insulin resistance in T2DM also occurs in platelets. As insulin directly inhibits platelet function, this mechanism might contribute to platelet activation and platelet hyperreactivity, which were in fact detected in diabetic patients. Since (inadvertent) platelet activation is causally linked to the development of atherosclerosis and atherothrombosis, regulation of platelet function is of utmost importance. Exercise training, performed on a regular basis has been shown to reduce morbidity and mortality in sedentary and diseased populations. Furthermore, exercise training improves whole body insulin sensitivity - however, it is currently unclear, if exercise training also affects insulin sensitivity of platelets. Recently, a time-saving interval training protocol has been adapted for T2DM-patients. Since this adapted high intensity interval training (HIIT) needs a fractional time commitment of exercise training according to current guidelines, HIIT possibly represents a promising instrument to increase adherence to exercise and thereby reduce T2DM morbidity.

Aims:

The primary aim of this study is to investigate the effect of 12 weeks of HIIT vs. continuous training (CT) on platelet insulin sensitivity and platelet (hyper)reactivity in prediabetic patients.

Secondary aims are to assess the effect of HIIT and CT on whole body insulin sensitivity and fitness in prediabetic patients as well as on various parameters of platelet function and on the hepatic fat content.

Hypotheses:

Our main hypothesis is that HIIT increases platelet insulin sensitivity and thereby decreases platelet activation/reactivity in patients with prediabetes. Methods: 44 prediabetic (see inclusion criteria) patients will be enrolled in this study. Patients will randomly be assigned to a HIIT group (committed to a supervised training program) or a CT group. After initial examinations (supervised graded exercise test, platelet function tests, oral glucose tolerance test, measurement of the hepatic fat content via FibroScan®), supervised training will be performed over a period of 12 weeks. Tests performed at the beginning of the study will be repeated after the training period.

ELIGIBILITY:
Inclusion Criteria:

* prediabetic (insulin-insensitive) patients
* either fasting plasma glucose 100- 125 mg/dl or HbA1c 5.7 - 6.4
* < 3kg bodyweight change within the last 6 months

Exclusion Criteria:

* Any contraindications for exercise
* resulting from anamnesis ( e.g. history of angina pectoris, peripheral arterial disease), ECG at rest or during graded exercise test, echocardiogram, echocardiography or lung function test
* chronical joint pain that makes exercise training on bicycle ergometers impossible
* any conditions that make the successful participation in the study unlikely
* islet cell autoantibodies
* Medication: insulin, thiazolidindiones, statins, antidepressants
* Secondary diseases: History of end-stage liver or kidney disease; pronounced neuropathy or retinopathy
* drug or alcohol abuse

Ages: 19 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2019-01-04 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2021-02 (Estimated)

PRIMARY OUTCOMES:
EC50 (half-maximal effective concentration) of TRAP-6 (thrombin-receptor activating peptide) in terms of surface CD62P (=platelet selectin, P-selectin) expression: group differences after 12 weeks of training | 12 weeks
EC50 of insulin in terms of intraplatelet VASP (vasodilator-stimulated phosphoprotein)-phosphorylation: group differences after 12 weeks of training | 12 weeks

SECONDARY OUTCOMES:
whole body insulin sensitivity | 12 weeks
Maximal oxygen consumption | 12 weeks
  Unit: ml/min/kg bodymass
EC50 of other platelet agonists in terms of various platelet activation markers | 12 weeks
EC50 of prostacyclin in terms of intraplatelet VASP-phosphorylation | 12 weeks
Transient elastography (FibroScan®) controlled attenuation parameter (CAP) | 12 weeks
  The controlled attenuation parameter (CAP) has demonstrated good accuracy in quantifying the levels of liver steatosis and fibrosis in patients with NAFLD
Fatty Liver Index (FLI) | 12 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- MUVienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: Undecided